CLINICAL TRIAL: NCT04534114
Title: Factor XI LICA to Reduce Thrombotic Events in End-Stage Renal Disease Patients on Hemodialysis: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of BAY 2976217
Brief Title: Factor XI LICA to Reduce Events Such as Heart Attack and Stroke in Patients Whose Kidneys Are no Longer Able to Work as They Should and Require Treatment to Filter Wastes From the Blood: Focus is on the Safety of BAY2976217 and the Way the Body Absorbs, Distributes and Removes the Study Drug
Acronym: RE-THINc ESRD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21170; 2019-003927-39 (EudraCT Number)
Record Dates: First submitted 2020-08-20; First posted 2020-09-01 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: End Stage Renal Disease Requiring Hemodialysis
Keywords: End stage renal disease (ESRD); Hemodialysis (HD); Thrombotic Events
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pooled Placebo (Placebo Comparator): Participants received subcutaneous treatment with matching placebo.
  Interventions: Drug: Placebo
- 40 mg BAY2976217 (Experimental): Participants received subcutaneous treatment with 40 mg BAY2976217.
  Interventions: Drug: Fesomersen sodium (BAY2976217)
- 80 mg BAY2976217 (Experimental): Participants received subcutaneous treatment with 80 mg BAY2976217.
  Interventions: Drug: Fesomersen sodium (BAY2976217)
- 120 mg BAY2976217 (Experimental): Participants received subcutaneous treatment with 120 mg BAY2976217.
  Interventions: Drug: Fesomersen sodium (BAY2976217)

INTERVENTIONS:
Drug: Fesomersen sodium (BAY2976217) — Study intervention will be injected subcutaneously.
  Other Names: Factor XI LICA
  Arms: 120 mg BAY2976217; 40 mg BAY2976217; 80 mg BAY2976217
Drug: Placebo — Matching placebo to BAY2976217 will be injected subcutaneously.
  Arms: Pooled Placebo

SUMMARY:
Patients whose kidneys are no longer able to work as they should and require treatment to filter wastes from the blood (hemodialysis) are at high risk for blood clots that form in blood vessels (thrombosis) blocking blood flow that causes heart attacks, strokes, and other life-threatening conditions. BAY2976217 is under clinical development for prevention of thrombosis. The goal of the study is to learn more about the safety of BAY2976217, how it is tolerated and the way the body absorbs, distributes and gets rid of the study dug given as multiple doses in participants with renal impairment who require hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years of age at the time of signing the informed consent form (ICF)
* Participants with ESRD on hemodialysis (HD) for ≥3 months at the time of signing of the ICF, receiving dialysis at least 9 hours a week and stable in the view of the investigator
* Male or female (contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies)
* Capable of giving signed ICF as described in the Protocol, which includes compliance with the requirements and restrictions listed in the ICF and in the protocol

Exclusion Criteria:

* Participants receiving antiplatelet therapy except daily acetylsalicylic acid (ASA) ≤ 150 mg/day
* Participants receiving anticoagulation in therapeutic doses, other than standard anticoagulation during the hemodialysis procedure
* Known inherited bleeding disorder e.g. von-Willebrand disease or Hemophilia A, B or C
* Recent (<6 months before screening) clinically significant bleeding, or at high risk of bleeding (in the judgement of the investigator)
* Recent (<3 months before screening) thromboembolic event, e.g. acute coronary syndrome, stroke, or Venous thromboembolism (except dialysis access thrombosis)
* Recent (<3 months before screening) major surgery or scheduled major surgery during participation in the study
* Scheduled living donor renal transplant during study participation
* Known Hepatitis B or C
* Known HIV with recent documented detectable viral load (<3 months before screening)
* Persistent heart failure as classified by the New York Heart Association classification of 3 or higher
* Life expectancy less than 6 months
* Sustained uncontrolled hypertension (persistent measurements of diastolic blood pressure ≥ 100 mmHg, and/or systolic blood pressure ≥ 180 mmHg)
* Hepatic disease associated with either: coagulopathy leading to a clinically relevant bleeding risk, or ALT > 3x ULN, or total bilirubin >2x ULN with direct bilirubin > 20% of the total
* Hb < 9.0 g/dL at screening
* Platelet count < 120,000 mm^3 at screening
* Known hypersensitivity to the investigational drug or to inactive constituents of the study intervention
* Active malignancy requiring treatment during study participation (except non-melanoma skin cancer, or cervical carcinoma in situ)
* Participation in a study with an investigational medicinal product within 30 days or within 5 half-lives of the previous administered drug, whichever is longer, prior to the screening/observational period (Note: Participants from previous BAY2306001/ISIS 416858 and BAY2976217/ ION 957943 studies are eligible)
* Any other conditions, which, in the opinion of the investigator or Sponsor would make the subject unsuitable for inclusion
* Confirmed pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (69):
- United States (9):
  - Fresenius Kidney Care Clovis, Clovis, California
  - Desert Cities Dialysis-Amethyst & Desert Cities Dialysis, Victorville, California
  - Davita East Ft. Lauderdale Dialysis Center, Fort Lauderdale, Florida
  - Fresenius Kidney Care St. Louis Regional Dialysis, Saint Ann, Missouri
  - Chromalloy Dialysis Center, St Louis, Missouri
  - Fresenius Medical Care - Fire Mesa Dialysis Unit, Las Vegas, Nevada
  - DaVita Northwest Medical Center Dialysis, San Antonio, Texas
  - San Antonio Kidney Disease Center Physicians Group, PLLC, San Antonio, Texas
  - Salem VA Medical Center, Salem, Virginia
- Belgium (4):
  - OL Vrouwziekenhuis - Campus Aalst, Aalst
  - UZ Brussel, Bruxelles - Brussel
  - UZ Antwerpen, Edegem
  - Regionaal ZH Jan Yperman Campus Mariaziekenhuis, Ieper
- Bulgaria (4):
  - First Dialysis Services Bulgaria Ead, Montana
  - MHAT Samokov, Samokov
  - MHAT "Knyaginya Klementina - Sofia"EAD, Sofia
  - MHAT National Cardiology Hospital EAD, Sofia
- Canada (6):
  - Etobicoke General Hospital, Etobicoke, Ontario
  - St. Joseph's Healthcare - Hamilton, Hamilton, Ontario
  - Lakeridge Health-Oshawa, Oshawa, Ontario
  - Unity Health Toronto: St. Michael's Hospital, Toronto, Ontario
  - Centre de services ambulatoires de dialyse de Gaspé, Montreal, Quebec
  - CHU de Québec-Université Laval, Québec
- Czechia (4):
  - Nemocnice Frydek-Mistek, Frýdek-Místek
  - Klatovska nemocnice, Klatovy
  - Fresenius Medical Care - DS, s.r.o., Mělník
  - Oblastni nemocnice Mlada Boleslav, Mladá Boleslav
- Germany (3):
  - DaVita Clinical Research Deutschland GmbH, Düsseldorf, North Rhine-Westphalia
  - DaVita Clinical Resarch Germany GmbH, Geilenkirchen, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein (UKSH), Kiel, Schleswig-Holstein
- Greece (3):
  - University General Hospital of Heraklion, Heraklion
  - University General Hospital of Patra, Pátrai
  - PAPANIKOLAOU General Hospital Thessaloniki, Pilea Chortiatis
- Hungary (2):
  - Bacs-Kiskun Megyei Korhaz, Kalocsa
  - SZTE ÁOK Szent Györgyi Albert Klinikai Kozpont, Szeged
- Japan (7):
  - Matsunami General Hospital, Hashima-gun, Gifu
  - Sapporo Tokushukai Hospital, Sapporo, Hokkaido
  - Ibaraki Prefectural Central Hospital, Kasama, Ibaraki
  - Public Central Hospital of Matto Ishikawa, Hakusan, Ishikawa-ken
  - Shonan Fujisawa Tokushukai Hospital, Fujisawa, Kanagawa
  - Hanyu General Hospital, Hanyū, Saitama
  - Medical corporation association Shunshin-kai Inage hospital, Chiba
- Latvia (4):
  - Daugavpils Regional Hospital, Daugavpils
  - Liepaja Regional Hospital, Liepāja
  - P. Stradins Clinical University Hospital, Riga
  - Vidzemes Hospital, Valmiera
- Russia (8):
  - High Technology Center Clinic 1, Moscow
  - Limited Liability Company "Nefroline-Novosibirsk", Novosibirsk
  - LLC Frezenius Nefrocare, Penza
  - LLC Dialysis center, Podolsk
  - Botkin clinical infectious diseases hospital, Saint Petersburg
  - LLC B. Brown Avitum Russland Clinics, Saint Petersburg
  - State Budgetary Healthcare Institution City Hospital #26, Saint Petersburg
  - Nikiforov All-Russian Center of Emergency and Radiation Med, Saint Petersburg
- South Korea (2):
  - The Catholic University of Korea, Incheon St.Mary's Hospital, Incheon, Incheon Gwang''yeogsi
  - Yeouido St. Mary's Hospital, Seoul, Seoul Teugbyeolsi
- Spain (5):
  - Hospital Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitari de Bellvitge | Bellvitge Biomedical Research Institute - Cardiology - AF, Stroke Prevention, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitario Virgen de las Nieves|Nefrologia, Granada
  - Hospital Universitari i Politècnic La Fe | Nefrología, Valencia
- Taiwan (2):
  - Chi Mei Medical Center, Tainan
  - Taipei Medical University Hospital, Taipei
- Ukraine (6):
  - Medical Center Fresenius Medical Care Ukraine, LLC, Chernihiv
  - Kyiv City Center of Nephrology and Dialysis, Kyiv
  - Kyiv Regional Clinical Hospital, Kyiv
  - Regional Clinical Hospital - Odessa, Odesa
  - Ternopil Regional Clinical Hospital, Ternopil
  - Zaporizhia Municipal Clinical Hospital No.10, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No
There are no current plans to share data. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Stamellou E, Noels H, Floege J. Factor XI inhibition in hemodialysis patients: the safer anticoagulation? Kidney Int. 2024 Jul;106(1):21-23. doi: 10.1016/j.kint.2024.03.029. PMID 38906653
- [Derived] Winkelmayer WC, Lensing AWA, Thadhani RI, Mahaffey KW, Walsh M, Pap AF, Willmann S, Thelen K, Hodge S, Solms A, Ingham SJM, Eikelboom J; RE-THINC investigators. A Phase II randomized controlled trial evaluated antithrombotic treatment with fesomersen in patients with kidney failure on hemodialysis. Kidney Int. 2024 Jul;106(1):145-153. doi: 10.1016/j.kint.2024.02.024. Epub 2024 Mar 26. PMID 38537676
- See also: Click here to find information about studies related to Bayer AG products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 69 study centers in 15 countries between 04-SEP-2020 (first participant first visit) and 12-MAY-2022 (last participant last visit).
Pre-assignment Details: From 359 participants screened, 51 participants were screening failure and a total of 308 participants were randomized and 307 were treated either with fesomersen or placebo.
Groups:
- Fesomersen 40 mg: Participants received monthly subcutaneous treatment with 40 mg fesomersen (Factor XI LICA). LICA=Ligand conjugated antisense oligonucleotide.
- Fesomersen 80 mg: Participants received monthly subcutaneous treatment with 80 mg fesomersen (Factor XI LICA). LICA=Ligand conjugated antisense oligonucleotide.
- Fesomersen 120 mg: Participants received monthly subcutaneous treatment with 120 mg fesomersen (Factor XI LICA). LICA=Ligand conjugated antisense oligonucleotide.
- Placebo: Participants received monthly subcutaneous treatment with matching placebo to fesomersen (Factor XI LICA). LICA=Ligand conjugated antisense oligonucleotide.
Period: Main Treatment Period
Arm/Group | Fesomersen 40 mg | Fesomersen 80 mg | Fesomersen 120 mg | Placebo
Started | 77 | 79 | 76 | 75
Completed | 67 | 66 | 64 | 61
Not Completed | 10 | 13 | 12 | 14
Not completed — COVID-19 pandemic: Participant decision | 0 | 1 | 0 | 0
Not completed — COVID-19 pandemic: Death | 0 | 1 | 0 | 2
Not completed — COVID-19 pandemic: Adverse event | 0 | 1 | 1 | 0
Not completed — COVID-19 pandemic: withdrawal following protocol | 1 | 3 | 3 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Death | 1 | 0 | 0 | 1
Not completed — Other reason | 1 | 1 | 0 | 0
Not completed — Participant decision | 1 | 3 | 3 | 1
Not completed — Protocol-specified withdrawal criterion met | 2 | 1 | 4 | 6
Not completed — Adverse Event | 4 | 2 | 1 | 2
Period: Extension Treatment Period
Arm/Group | Fesomersen 40 mg | Fesomersen 80 mg | Fesomersen 120 mg | Placebo
Started | 62 | 61 | 63 | 58
Completed | 59 | 57 | 62 | 53
Not Completed | 3 | 4 | 1 | 5
Not completed — COVID-19 pandemic: Death | 0 | 0 | 0 | 1
Not completed — COVID-19 pandemic: withdrawal following protocol | 1 | 0 | 0 | 0
Not completed — Other reason | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 1
Not completed — Protocol-specified Withdrawal Criterion Met | 2 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fesomersen 40 mg | Fesomersen 80 mg | Fesomersen 120 mg | Placebo | Total
Number analyzed (Participants) | 77 | 79 | 76 | 75 | 307
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (13.2) | 58.0 (14.4) | 57.7 (13.3) | 58.6 (11.9) | 58.7 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 20 | 30 | 22 | 107
  Male | 42 | 59 | 46 | 53 | 200
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 1 | 2 | 12
  Not Hispanic or Latino | 74 | 73 | 75 | 72 | 294
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 12 | 8 | 11 | 13 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 4 | 1 | 8
  White | 62 | 70 | 61 | 61 | 254
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Composite of Major Bleeding (MB) and Clinically-relevant Non-major Bleeding (CRNMB) During the Main Treatment Period and Within the On-treatment Time Window, as Assessed by Blinded Central Independent Adjudication Committee (CIAC)
Description: MB is defined as symptomatic bleeding and: 1) Fatal bleeding, and/or; 2) Bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome, and/or; 3) Bleeding causing a fall in hemoglobin level of 20 g/L (2.0 g/dL) (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells. CRNMB is defined as any sign or symptom of hemorrhage that does not fit the criteria for the ISTH definition of major bleeding but does meet at least one of the following criteria: 1) Requiring medical intervention by a healthcare professional; 2) Leading to hospitalization or increased level of care; 3) Prompting a face-to-face evaluation. n/100 person-years: number of subjects with incident events divided by the cumulative at-risk time in the reference population, where a subject is no longer at risk once an incident event occurred.
Time Frame: Up to 24 weeks
Population: Safety analysis set (SAF) includes all randomized participants who received at least one dose of the study intervention according to actual treatment arm received.
Measure: Number (95% Confidence Interval); unit: n/100 person-years
Arm/Group | Fesomersen 40 mg | Fesomersen 80 mg | Fesomersen 120 mg | Placebo
Number analyzed (Participants) | 77 | 79 | 76 | 75
n/100 person-years | 9.0 [2.5 to 18.9] | 9.1 [2.5 to 19.1] | 6.1 [1.1 to 14.5] | 9.7 [2.7 to 20.4]
Statistical Analysis 1: Comparison: Fesomersen 40 mg vs Placebo; Test type: Other — Fesomersen groups were compared to the placebo group using two-sided log-rank tests. Due to the exploratory nature of these analyses, no multiplicity adjustment was done. Cause-specific hazard ratio and corresponding 2-sided 95% confidence intervals, comparing the hazards for the event-of-interest in each of the Fesomersen groups with the placebo group were estimated based on three separate cause-specific Cox proportional hazards models as exploratory analysis; p = 0.944, Log Rank; Cause specific Hazard ratio = 0.94, 95% CI 2-sided [0.19 to 4.68]
Statistical Analysis 2: Comparison: Fesomersen 80 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.953, Log Rank; Cause specific Hazard ratio = 0.95, 95% CI 2-sided [0.19 to 4.72]
Statistical Analysis 3: Comparison: Fesomersen 120 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.605, Log Rank; Cause specific Hazard ratio = 0.63, 95% CI 2-sided [0.10 to 3.75]

2. Secondary Outcome: Incidence of Composite of MB and CRNMB During the Main and Extended Treatment Periods and Within the On-treatment Time Window, as Assessed by Blinded CIAC
Description: as for outcome 1
Time Frame: Up to 48 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: n/100 person-years
Arm/Group | Fesomersen 40 mg | Fesomersen 80 mg | Fesomersen 120 mg | Placebo
Number analyzed (Participants) | 77 | 79 | 76 | 75
n/100 person-years | 10.7 [4.2 to 19.7] | 8.6 [2.9 to 16.7] | 6.4 [1.7 to 13.3] | 7.0 [1.9 to 14.8]
Statistical Analysis 1: Comparison: Fesomersen 40 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.612, Log Rank; Cause specific Hazard ratio = 1.45, 95% CI 2-sided [0.34 to 6.08]
Statistical Analysis 2: Comparison: Fesomersen 80 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.757, Log Rank; Cause specific Hazard ratio = 1.27, 95% CI 2-sided [0.28 to 5.66]
Statistical Analysis 3: Comparison: Fesomersen 120 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.909, Log Rank; Cause specific Hazard ratio = 0.91, 95% CI 2-sided [0.18 to 4.52]

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) During the Main Treatment Period and Within the On-treatment Time Window and Their Severity
Description: TEAEs were analyzed during the on-treatment time window within the main treatment period in the safety analysis set (SAF). Data observed from the randomization date until the end of the main treatment period. TEAEs were defined as events occurring after first study intervention administration and up to 20 weeks after last study intervention administration.
Time Frame: Up to 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fesomersen 40 mg | Fesomersen 80 mg | Fesomersen 120 mg | Placebo
Number analyzed (Participants) | 77 | 79 | 76 | 75
Participants
  Any TEAE | 54 | 56 | 55 | 55
  Maximum intensity for any TEAE: Mild | 28 | 28 | 22 | 27
  Maximum intensity for any TEAE: Moderate | 17 | 24 | 28 | 19
  Maximum intensity for any TEAE: Severe | 9 | 4 | 5 | 9

4. Secondary Outcome: Number of Participants With TEAEs During the Main and Extended Treatment Periods and Within the On-treatment Time Window and Their Severity
Description: TEAEs were analyzed during during main and extended treatment periods in the safety analysis set (SAF). Data observed from the randomization date until the end of the extension treatment period. TEAEs were defined as events occurring after first study intervention administration and up to 20 weeks after last study intervention administration.
Time Frame: Up to 48 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fesomersen 40 mg | Fesomersen 80 mg | Fesomersen 120 mg | Placebo
Number analyzed (Participants) | 77 | 79 | 76 | 75
Participants
  Any TEAE | 61 | 62 | 58 | 56
  Maximum intensity for any TEAE: Mild | 26 | 25 | 20 | 26
  Maximum intensity for any TEAE: Moderate | 24 | 31 | 30 | 18
  Maximum intensity for any TEAE: Severe | 11 | 6 | 8 | 12

5. Secondary Outcome: Number of Participants With TEAEs During the Main and Extended Treatment Periods and Until 20 Weeks After the Last Study Intervention Dose and Their Severity
Description: TEAEs occurring from first study intervention intake until 20 weeks after last study intervention intake.
Time Frame: Up to 48 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fesomersen 40 mg | Fesomersen 80 mg | Fesomersen 120 mg | Placebo
Number analyzed (Participants) | 77 | 79 | 76 | 75
Participants
  Any TEAE | 64 | 63 | 62 | 59
  Maximum intensity for any TEAE: Mild | 21 | 21 | 18 | 21
  Maximum intensity for any TEAE: Moderate | 28 | 33 | 33 | 22
  Maximum intensity for any TEAE: Severe | 15 | 9 | 11 | 16

6. Secondary Outcome: Trough Concentrations (Ctrough) of Three Dose Levels of Fesomersen
Description: Trough (pre-dose) fesomersen-equivalent plasma concentrations (Ctrough) for 3 dose levels of fesomersen were summarized descriptively by dose level and visit: Visit 12, Visit 14, Visit 16, Visit 18 (main treatment period). Ctrough was not measured for the placebo group.
Time Frame: At visits V12 (Day 57), V14 (Day 85), V16 (Day 113), V18 (Day 141)
Population: Pharmacokinetic analysis set (PKS) includes all fesomersen-treated participants with at least 1 PK sample in accordance with the PK sampling schedule and without deviation from the protocol that would interfere with the evaluation of the PK data were included in the PK analysis. Only those participants who have sample collection with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Fesomersen 40 mg | Fesomersen 80 mg | Fesomersen 120 mg
Number analyzed (Participants) | 77 | 79 | 76
μg/mL
  Visit 12: number analyzed (Participants) | 62 | 57 | 55
  Visit 12 | 0.000454 (118.753791) | 0.000704 (80.938271) | 0.001186 (76.691406)
  Visit 14: number analyzed (Participants) | 62 | 60 | 62
  Visit 14 | 0.000490 (92.511801) | 0.000792 (82.170296) | 0.001246 (97.530820)
  Visit 16: number analyzed (Participants) | 58 | 56 | 60
  Visit 16 | 0.000572 (85.974878) | 0.000789 (68.188121) | 0.001346 (81.805680)
  Visit 18: number analyzed (Participants) | 64 | 53 | 59
  Visit 18 | 0.000521 (106.848825) | 0.000828 (91.024162) | 0.001424 (92.709743)

7. Secondary Outcome: Maximum Change in FXI (Coagulation Factor XI) Antigen Levels During the Main Treatment Period
Description: The secondary endpoint of change in FXI antigen levels during the main treatment period was an optional secondary endpoint only as mentioned in the integrated clinical protocol amendment version 3.0 and was not analyzed in this study as the FXI activity assay is sufficient to describe the effect on FXI level in plasma.
Time Frame: Up to 24 weeks
Population: Pharmacodynamic set (PDS) includes all participants with at least 1 PD sample in accordance with the PD sampling schedule and without deviation from the protocol that would interfere with the evaluation of the PD data were included in the PD analysis. Data were not collected for this outcome measure.
Arm/Group | Fesomersen 40 mg | Fesomersen 80 mg | Fesomersen 120 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Maximum Change in FXI Activity Levels During the Main Treatment Period
Description: The FXIa activity was measured by a fluorogenic activated FXIa activity (AXIA) assay. Absolute change from baseline at each visit until Visit 22 (Day 169) are reported.
Time Frame: Baseline, Days 1 (Pre-Dose and 5 hours post-dose), 2, 8, 15, 22, 29 (Pre-dose and 5 hours post-dose), 43, 57 (Pre-dose), 71, 85 (Pre-dose), 113 (Pre-dose), 141 (Pre-dose),148, 155, 162, and 169 (Pre-dose)
Population: Pharmacodynamic set (PDS) includes all participants with at least 1 PD sample in accordance with the PD sampling schedule and without deviation from the protocol that would interfere with the evaluation of the PD data were included in the PD analysis.
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Fesomersen 40 mg | Fesomersen 80 mg | Fesomersen 120 mg | Placebo
Number analyzed (Participants) | 77 | 79 | 76 | 75
U/mL
  Baseline | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Visit 5 (Day 1): Pre-dose | 0.06 (0.06) | 0.05 (0.06) | 0.05 (0.05) | 0.04 (0.05)
  Visit 5 (Day 1): 5 Hours | 0.09 (0.09) | 0.11 (0.12) | 0.13 (0.13) | 0.10 (0.08)
  Visit 6 (Day 2): 22 Hours | 0.13 (0.11) | 0.12 (0.12) | 0.15 (0.13) | 0.14 (0.13)
  Visit 7 (Day 8) | 0.21 (0.15) | 0.32 (0.15) | 0.43 (0.18) | 0.08 (0.07)
  Visit 8 (Day 15) | 0.34 (0.23) | 0.48 (0.21) | 0.61 (0.24) | 0.12 (0.09)
  Visit 9 (Day 22) | 0.37 (0.26) | 0.50 (0.23) | 0.63 (0.25) | 0.11 (0.09)
  Visit 10 (Day 29): Pre-dose | 0.34 (0.26) | 0.44 (0.21) | 0.60 (0.25) | 0.09 (0.07)
  Visit 10 (Day 29): 5 Hours | 0.32 (0.25) | 0.43 (0.22) | 0.58 (0.25) | 0.12 (0.14)
  Visit 11 (Day 43) | 0.47 (0.29) | 0.59 (0.25) | 0.76 (0.27) | 0.09 (0.08)
  Visit 12 (Day 57): Pre-dose | 0.42 (0.26) | 0.55 (0.24) | 0.69 (0.28) | 0.11 (0.10)
  Visit 13 (Day 71) | 0.52 (0.26) | 0.66 (0.24) | 0.76 (0.25) | 0.15 (0.13)
  Visit 14 (Day 85): Pre-dose | 0.46 (0.27) | 0.59 (0.26) | 0.72 (0.24) | 0.14 (0.12)
  Visit 16 (Day 113): Pre-dose | 0.46 (0.26) | 0.57 (0.28) | 0.75 (0.25) | 0.16 (0.16)
  Visit 18 (Day 141): Pre-dose | 0.47 (0.27) | 0.56 (0.28) | 0.72 (0.25) | 0.12 (0.09)
  Visit 19 (Day 148) | 0.52 (0.27) | 0.63 (0.29) | 0.76 (0.26) | 0.15 (0.16)
  Visit 20 (Day 155) | 0.52 (0.28) | 0.65 (0.29) | 0.77 (0.25) | 0.15 (0.17)
  Visit 21 (Day 162) | 0.50 (0.30) | 0.64 (0.28) | 0.75 (0.26) | 0.16 (0.20)
  Visit 22 (Day 169): Pre-dose | 0.46 (0.29) | 0.59 (0.28) | 0.73 (0.25) | 0.17 (0.21)

ADVERSE EVENTS:
Time Frame: From first study intervention up to 64 Weeks.
Description: Adverse event reporting for the all-cause mortality considers all deaths that occurred at any time during the study before the last contact, up to 64 Weeks.
Arm/Group | Fesomersen 40 mg | Fesomersen 80 mg | Fesomersen 120 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 2/77 | 1/79 | 2/76 | 7/75
Serious Adverse Events (participants affected / at risk) | 19/77 | 18/79 | 17/76 | 20/75
Other Adverse Events (participants affected / at risk) | 31/77 | 27/79 | 30/76 | 21/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fesomersen 40 mg (N=77) | Fesomersen 80 mg (N=79) | Fesomersen 120 mg (N=76) | Placebo (N=75)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spleen ischaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic ischaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular access site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 4 (4) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 4 (4) | 1 (1) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 3 (7)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shunt occlusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shunt stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delayed graft function (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous graft site pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transplant evaluation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Klebsiella test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post cardiac arrest syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal transplant (Surgical and medical procedures) | 3 (3) | 4 (4) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fesomersen 40 mg (N=77) | Fesomersen 80 mg (N=79) | Fesomersen 120 mg (N=76) | Placebo (N=75)
Anaemia (Blood and lymphatic system disorders) | 4 (6) | 4 (9) | 3 (5) | 4 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (5) | 7 (13) | 7 (11) | 2 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (9) | 2 (2) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 7 (8) | 3 (4) | 2 (3) | 4 (4)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 4 (4) | 2 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (10) | 3 (5) | 5 (7) | 3 (13)
Headache (Nervous system disorders) | 4 (4) | 3 (4) | 3 (5) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (3) | 4 (4) | 3 (3) | 2 (3)
Hypertension (Vascular disorders) | 3 (5) | 5 (9) | 6 (8) | 7 (8)
Hypotension (Vascular disorders) | 6 (27) | 4 (12) | 8 (12) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study may be published or presented at scientific meetings. If this is foreseen, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission. This allows the sponsor to protect proprietary information and to provide comments.

DOCUMENTS (2):
  • Study Protocol (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT04534114/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/14/NCT04534114/SAP_001.pdf